CLINICAL TRIAL: NCT04564651
Title: Platelet Transfusion in Acute-on Chronic Liver Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Jinjun Chen, Associate Director, Nanfang Hospital, Southern Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 013
Record Dates: First submitted 2020-09-18; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Platelet Transfusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- platelet transfusion treatment (Experimental)
  Interventions: Other: platelet transfusion
- standard medical treatment (No Intervention)

INTERVENTIONS:
Other: platelet transfusion — when the ADP inhibition >70%, give one unit platelet tansfusion
  Arms: platelet transfusion treatment

SUMMARY:
Acute on-chronic liver failure (ACLF) is a severe liver disease with a 28-day mortality rate of up to 40%. When the patients get 3 or more organ failures, the 28-day mortality rate is up to 82.6%. Though the ACLF patients have high short-term mortality, and the only effective treatment method is liver transplantation. However, few patients can be treated due to the scarcity of liver source, rapid disease progression and short transplantation window.

Our team evaluated the platelet function of 100 patients with ACLF by using the thromboelastograghy (TEG 5000). It was found for the first time that the reactivity of platelets of ACLF patients decreased, and the platelet inhibition rate (especially the ADP pathway) was related to patients'short-term prognosis. When the ADP inhibition rate was 70%, the patients'28-day mortality was up to 100%. However, the mechanism of low platelet response to ADP in ACLF patients is still unclear. We found that the platelet function in patients with ACLF 2-3 grade and inhibition rate beyond 70% was improved and the 28-day mortality decreased after platelet transfusion. Whether platelet transfusion can prolong survival time needs to be determined in a prospective controlled study. Therefore, this study is expected to find a new therapeutic method to reduce the mortality of patients with ACLF.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old;
* Patients with compensated cirrhosis conformed to the (ACLF) diagnostic criteria of chronic and acute liver failure defined by the European Association of Hepatology (EASL-CLIF), and met the ACLF-2 and 3 grades.

ADP inhibition rate ≥ 70%.

Exclusion Criteria:

* Patients with severe platelet allergy in the past;
* Coma caused by cerebral hemorrhage or primary diseases of the nervous system;
* Those who have taken anti-platelet drugs or anticoagulants within four weeks;
* Rupture and bleeding of EVB occurred within 1 week.
* Those who received platelet transfusion within 1 week;
* Patients with liver cancer or other malignant tumors;
* Pregnant and lactating women;
* Complicated with other serious chronic diseases;
* Not signing the informed consent form;
* Other researchers do not consider it appropriate to participate in the study.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
28-day transplant-free mortality | 28 days
  whether participant died or not without liver transplantation

SECONDARY OUTCOMES:
90-day transplant-free mortality | 90 days
  mortality without transplant in 90 day

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - The First Affiliated Hospital of Army Medical University, Chongqing, Chongqing Municipality
  - Nanfang Hospital, Guangzhou, Guangdong
  - Taihe Hospital affiliated to Hubei Medical College, Shiyan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Xinjiang Medical University, Xinjiang, Xinjiang
  - Meng Chao Hepatobiliary Hospital of Fujian Medical University, Fujian
  - Shanghai Public Health Clinical Center, Shanghai

IPD SHARING:
Plan to Share IPD: No